CLINICAL TRIAL: NCT07101991
Title: Effects of Goal-directed Fluid Management Guided by a Non-invasive Device on the Incidence of Postoperative Complications in Neurosurgery: a Multicenter, Prospective, Randomized, Controlled Study
Brief Title: Effects of GDHT (Goal Directed Hemodynamic Therapy) Using a Non-invasive Hemodynamic Monitoring in Elective Neurosurgery
Acronym: NCHGDT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brno University Hospital (Other)
Collaborators: Military University Hospital, Prague (Other); Zlin Regional Hospital (Unknown)
Responsible Party: Principal Investigator, Roman Gal, Head of the department, Brno University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT0012025
Record Dates: First submitted 2025-07-03; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Surgery Complications
Keywords: neurosurgery; goal-directed therapy; adverse events
MeSH Terms: interventions — Early Goal-Directed Therapy

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard monitoring (Active Comparator): In this arm standard monitoring of vital signs will be used during operation.
  Interventions: Other: Standard monitoring
- Goal-Directed Therapy (Experimental): A non-invasive hemodynamic monitor STARLINK™SV will be used in addition to standard monitoring.
  Interventions: Other: Goal-Directed Therapy

INTERVENTIONS:
Other: Standard monitoring — Administration of fluids and vasoactive drugs guided by standard vital signs monitoring
  Arms: Standard monitoring
Other: Goal-Directed Therapy — Administration of fluids and vasoactive drugs guided by non-invasive haemodynamic monitoring
  Arms: Goal-Directed Therapy

SUMMARY:
This study aims to assess the safety and efficacy of GDHT using the non-invasive Starling™ SV System in elective neurosurgery. The tested group of patients (n=70) will be compared with a control group (n=70), where hemodynamic management will be guided by standard vital signs monitoring.

DETAILED DESCRIPTION:
Patients undergoing major surgery are at risk for inadequate intravascular volumes and therefore inadequate tissue perfusion and oxygen delivery. Especially in neurosurgery, fluid management can be a challenge. In many surgical areas, such as orthopedics, gynecology or abdominal surgery, goal-directed fluid therapy is used with the aim of reducing postoperative complications. Current knowledge regarding effect of the goal-directed therapy in neurosurgery is limited.

This is a multicenter, prospective, randomized, controlled study that compares two approaches to fluid management in elective brain surgery. Patients scheduled for brain surgery will be screened whether they meet the inclusion criteria and after obtaining informed consent, the patient will be randomized to one of two study arms.

In the first (standard) arm standard vital signs monitoring will be used during the surgery and perioperative fluid management and administration of vasopressors will be guided by the decision of the attending anaesthetist.

In the second (GDT) arm perioperative fluid management and administration of vasopressors will be guided by a non-invasive hemodynamic monitor STARLINK™SV, which will be introduced in addition to standard monitoring.

The primary outcome is the incidence of adverse events and reactions according to following Adverse Events of Special Interest (AESI) in both study groups and their comparison. The secondary outcome is to investigate the efficacy and additional safety parameters of GDHT guided by non-invasive advanced hemodynamic monitoring versus hemodynamic management guided by standard vital signs monitoring.

This study will enroll 140 patients in total, 70 in each group. After completion of enrolment of patients the statistical analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for the trial if they meet all of the following criteria:

* Age ≥ 18 years
* Elective brain surgery with an expected duration ≥ 2 h
* Category 1-3 according to the ASA (American Society of Anesthesiologists) Physical Status Classification
* Lateral or supine operative position
* Signed the relevant informed consent form

Exclusion Criteria:

Subjects will not be eligible for the trial if they meet any of the following criteria:

* Category 4 according to the ASA Physical Status Classification
* Surgery for traumatic brain injury or acute hemorrhagic stroke
* Awake brain surgery
* Osmotherapy before surgery (with the exception of prophylactic administration of osmotic agents according to institutional standards)
* Unavailability of hemodynamic monitoring data
* Cardiac arrhythmia with irregular cardiac rhythm
* Known hypersensitivity to the active substance or to any of the excipients of IMP (Investigational Medicinal Product)
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with acute kidney Injury | 28 days
  Defined according to Kidney Disease Improving Global Outcomes (KDIGO) guidelines: Stage 1: serum creatinine 1.5-1.9 times baseline value within 7 days or ≥27 µmol l-1 (0.3 mg dl-1) increase within 48 h; urine output ≤0.5 ml kg-1 h-1 for 6-12 h Stage 2: serum creatinine 2.0-2.9 times baseline value within 7 days; urine output ≤0.5 ml kg-1 h-1 for 12 h Stage 3: serum creatinine 3.0 times baseline within 7 days or increase in serum creatinine to ≥354 µmol l-1 (≥4.0 mg.dl1 with an acute rise of > 44 mmol l-1 (0.5 mg/dl-1) or initiation of renal replacement therapy or in patients < 18 years, decrease in eGFR (estimated Glomerular Filtration Rate) to < 35 ml min-1 per 1.73m2; urine output ≤0.3 ml kg1 h-1 for 24 h or anuria for 12 h.
  AESI will be analysed descriptively and compared between study groups.
Number of participants with acute Respiratory Distress Syndrome (ARDS) | 28 days
  The Berlin definition of Respiratory Distress Syndrome:
  Timing: Within one week of a known clinical insult or new or worsening respiratory symptoms and Chest imaging: Bilateral opacities not fully explained by effusions, lobar/lung collapse or nobles and Origin of oedema: Respiratory failure not fully explained by cardiac failure or fluid overload.
  Need objective assessment (e.g. echocardiography) to exclude hydrostatic oedema if no risk factor is presented and Oxygenation disorder: mild: PaO2 (partial pressure of oxygen in arterial blood):FIO2 (Fraction of Inspired Oxygen) between 26.7 and 40.0 kPa (kilopascal) (200-300mmHg) with PEEP (Positive End-Expiratory Pressure) or CPAP (Continuous Positive Airway Pressure) ≥5 cmH2O (centimeters of water). Moderate: PaO2:FIO2 between 13.3 and 26.6 kPa (100- 200 mmHg) with PEEP ≥5 cmH2O. Severe: PaO2:FIO2 ≤13.3 kPa (100mmHg) with PEEP ≥5 cmH2O.
  AESI will be analysed descriptively and compared between study groups.
Number of participants with arrhythmia | 28 days
  Defined as electrocardiograph (ECG) evidence of cardiac rhythm disturbance. AESI will be analysed descriptively and compared between study groups.
Number of participants with cardiac arrest | 28 days
  Cessation of cardiac mechanical activity, as confirmed by the absence of signs of circulation. AESI will be analysed descriptively and compared between study groups.
Number of participants with cardiogenic pulmonary oedema | 28 days
  Defined as evidence of fluid accumulation in the alveoli due to poor cardiac function.
  AESI will be analysed descriptively and compared between study groups.
Number of participants with deep vein thrombosis (DVT) | 28 days
  A new blood clot or thrombus within the venous system. Appropriate diagnostic tests include ultrasound, venography, CT or MRI venography. Plasma D-dimer measurement is not recommended as a diagnostic test in the first three weeks following surgery.
  AESI will be analysed descriptively and compared between study groups.
Number of participants with pulmonary embolism (PE) | 28 days
  A new blood clot or thrombus within the pulmonary arterial system. AESI will be analysed descriptively and compared between study groups.
Number of participants with gastrointestinal bleed | 28 days
  Clinical or endoscopic evidence of blood in the gastrointestinal tract. AESI will be analysed descriptively and compared between study groups.
Number of participants with infection, source uncertain | 28 days
  Infection where there is strong clinical suspicion of infection but the source has not been confirmed because clinical information suggests more than one possible site, meeting two or more of the following criteria: core temperature < 36°C or >38°C; white cell count >12×109 l-1 or < 4×109 l-1, respiratory rate >20 breaths per minute or PaCO2 < 4.7 kPa (35mmHg); pulse rate >90 beats per minute.
  AESI will be analysed descriptively and compared between study groups.
Number of participants with laboratory confirmed bloodstream infection | 28 days
  Infection which meets at least one of the following criteria which should not be related to infection at another site:
  1. Patient has a recognised pathogen cultured from one or more blood cultures and the organism cultured from blood is not related to an infection at another site.
  2. Patient has at least one of the following signs or symptoms: fever >38°C, chills or hypotension, and at least one of the following.
     1. Common skin contaminant cultured from two or more blood cultures drawn on separate occasions.
     2. Common skin contaminant cultured from at least one blood culture from a patient with an intravascular line, and the physician institutes appropriate antimicrobial therapy.
     3. Positive blood antigen test. AESI will be analysed descriptively and compared between study groups.
Number of participants with myocardial infarction | 28 days
  Defined as increase in serum cardiac biomarker values (preferably cardiac troponin) with at least one value above the 99th percentile upper reference limit and at least one of the following criteria: symptoms of ischaemia; new or presumed new significant ST segment or T wave ECG changes or new left bundle branch block; development of pathological Q waves on ECG; radiological or echocardiographic evidence of new loss of viable myocardium or new regional wall motion abnormality; identification of an intracoronary thrombus at angiography or autopsy.
  AESI will be analysed descriptively and compared between study groups.
Number of participants with pneumonia | 28 days
  Definition: Two or more serial chest radiographs with at least one of the following (one radiograph is sufficient for patients with no underlying pulmonary or cardiac disease):
  1. new or progressive and persistent infiltrates
  2. consolidation
  3. cavitation; at least one of the following:
  (1) fever (>38°C) with no other recognised cause (2) leucopaenia (white cell count < 4 × 109 l-1) or leucocytosis (white cell count >12 × 109 l-1) (3) for adults >70 years old, altered mental status with no other recognised cause; and at least two of the following:
  1. new onset of purulent sputum or change in character of sputum, or increased respiratory secretions, or increased suctioning requirements
  2. new onset or worsening cough, or dyspnoea, or tachypnoea
  3. rales or bronchial breath sounds
  4. worsening gas exchange (hypoxaemia, increased oxygen requirement, increased ventilator demand).
  AESI will be analysed descriptively and compared between study groups.
Number of participants with paralytic ileus | 28 days
  Failure to tolerate solid food or defecate for three or more days after surgery.
  AESI will be analysed descriptively and compared between study groups.
Number of participants with postoperative haemorrhage | 28 days
  Blood loss within 72 h after the start of surgery which would normally result in transfusion of blood.
  AESI will be analysed descriptively and compared between study groups.
Number of participants with stroke | 28 days
  An embolic, thrombotic or haemorrhagic cerebral event with persistent residual motor, sensory or cognitive dysfunction (e.g. hemiplegia, hemiparesis, aphasia, sensory deficit, impaired memory).
  AESI will be analysed descriptively and compared between study groups.
Number of participants with brain oedema | 28 days
  Brain oedema confirmed on CT or MRI scan. AESI will be analysed descriptively and compared between study groups.
Number of participants with surgical site infection (superficial) | 28 days
  A superficial incisional surgical site infection is defined as one which meets the following criteria:
  1. Infection occurs within 30 days after surgery and
  2. Involves only skin and subcutaneous tissue of the incision and
  3. The patient has at least one of the following:
     1. purulent drainage from the superficial incision
     2. organisms isolated from an aseptically obtained culture of fluid or tissue from the superficial incision
     3. at least one of the following symptoms or signs of infection: pain or tenderness, localised swelling, redness or heat, and superficial incision is deliberately opened by surgeon and is culture positive or not cultured. A culture-negative finding does not meet this criterion.
     4. diagnosis of an incisional surgical site infection by a surgeon or attending physician.
  AESI will be analysed descriptively and compared between study groups.
Number of participants with surgical site infection (deep) | 28 days
  1. Infection occurs within 30 days after surgery if no implant is left in place or 1 year if implant is in place.
  2. Involves deep soft tissues (e.g. fascial and muscle layers) of the incision.
  3. The patient has at least one of the following:
     1. purulent drainage from the deep incision but not from the organ/space component of the surgical site
     2. a deep incision spontaneously dehisces or is deliberately opened by a surgeon and is culture-positive or not cultured when the patient has at least one of the following symptoms or signs: fever (>38°C), or localised pain or tenderness. A culture- negative finding does not meet this criterion.
     3. an abscess or other evidence of infection involving the deep incision is found on direct examination, during surgery, or by histopathological or radiological examination
     4. diagnosis of an incisional surgical site infection by a surgeon or attending physician.
  AESI will be analysed descriptively and compared between study groups.
Number of participants with surgical site infection (organ/space) | 28 days
  Infection which involves any part of the body excluding the fascia or muscle layers and meets the following criteria:
  1. Infection occurs within 30 days after surgery.
  2. The infection appears to be related to the surgical procedure and involves any part of the body, excluding the skin incision, fascia or muscle layers opened or manipulated during the operative procedure.
  3. The patient has at least one of the following:
     1. purulent drainage from a drain that is placed through a stab wound into the organ/space
     2. organisms isolated from an aseptically obtained culture of fluid or tissue in the organ/space
     3. an abscess or other evidence of infection involving the organ/space that is found on direct examination, during reoperation or by histopathological or radiological examination
     4. diagnosis of an organ/space surgical site infection by a surgeon or attending physician. AESI will be analysed descriptively and compared between study groups.
Number of participants with urinary tract infection | 28 days
  A positive urine culture of ≥105 colony forming units ml-1 with no more than two species of micro-organisms, and with at least one of the following symptoms or signs: fever (>38°C), urgency, frequency, dysuria, suprapubic tenderness, costovertebral angle pain or tenderness with no other recognised cause. Each of these criteria should be identified within a 24-h period.
  AESI will be analysed descriptively and compared between study groups.

SECONDARY OUTCOMES:
Duration of surgery | During the surgery (hours)
  Duration of surgery (min) - will be analysed descriptively and compared between study arms
Length of hospital stay | Days (up to 28)
  LOS (Length of stay, day of admission - day of discharge will be counted as 1 day) - will be calculated as a number of days between admission and discharge, analysed descriptively and compared between study groups.
ICU length of stay | Days (up to 28)
  ICU LOS (day of admission - day of discharge will be counted as 1 day) - will be calculated as a number of days between admission to the ICU and discharge from the ICU, analysed descriptively and compared between study groups.
28-day mortality | 28 days after randomization
  28-day mortality (number of patients who are not alive 28 days after randomization) will be evaluated as a number and percentage of patients who are not alive 28 days after randomization and compared between study arms.
Adverse events | 28 days
  Descriptive analysis of the incidence of any adverse events and reactions
Hemodynamic characteristics - MAP (Mean arterial pressure) | During the surgery and 24 hours post operation
  MAP (mmHg; before, after surgery) will be analysed descriptively and compared between study arms.
Hemodynamic characteristics - HR (Heart rate) | During the surgery and 24 hours post operation
  HR (Bpm; before, after surgery) will be analysed descriptively and compared between study arms.
Hemodynamic characteristics - SVV (Stroke volume variation) measured by The Starling™ SV System | During the surgery (hours)
  SVV (%; before, after surgery will be analysed descriptively and compared between study arms.
Hemodynamic characteristics - number of episodes of hypotension | During the surgery and 24 hours post operation
  Number of episodes of hypotension will be analysed descriptively and compared between study arms.
Hemodynamic characteristics - number of vasopressor administrations | During the surgery and 24 hours post operation
  Number of vasopressor administrations will be analysed descriptively and compared between study arms.
Hemoglobin | 24 hours
  Hemoglobin (g/l; before, after surgery and 24 hours after surgery) - will be analysed descriptively and compared between study arms.
Plasma lactate level | 24 hours
  Plasma lactate level (mmol/L; before, after surgery and 24 hours after surgery) will be analysed descriptively and compared between study arms.
Volume of blood loss | During the surgery and 24 hours post operation
  Volume of blood loss (ml/kg; during surgery and in the 24-hour postoperative period) will be analysed descriptively and compared between study arms.
Urinary output | During the surgery and 24 hours post operation
  Urinary output (ml/kg/hod; during surgery and in the 24-hour postoperative period) will be analysed descriptively and compared between study arms.
Number of administered units of packed RBC (Red blood cell) | During the surgery and 24 hours post operation
  Number of administered units of packed RBC (during surgery and in the 24-hour postoperative period) will be analysed descriptively and compared between study arms.
Number of subjects receiving transfusion | During the surgery and 24 hours post operation
  Number of subjects receiving transfusion (during surgery and in the 24-hour postoperative period) will be analysed descriptively and compared between study arms.
Crystalloid and colloid solutions consumption | During the surgery and 24 hours post operation
  Crystalloid and colloid solutions consumption (type and total volume of infusion during surgery and in the 24-hour postoperative period) will be analysed descriptively and compared between study arms.
Boluses of crystalloids | During the surgery and 24 hours post operation
  Boluses of crystalloids (ml; during surgery) will be analysed descriptively and compared between study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Veronika Kočí, M.D., Study Chair — The University Hospital Brno

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-05-29): https://cdn.clinicaltrials.gov/large-docs/91/NCT07101991/Prot_000.pdf